CLINICAL TRIAL: NCT01981213
Title: Attempted Suicide With Acetaminophen Among 8-18 Year-old Children / Adolescents
Brief Title: Attempted Suicide With Acetaminophen Among 8-18 Year-old Children / Adolescents in Denmark
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillerod Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Rikke Hedeland, MD, Hillerod Hospital, Denmark
Other Study IDs: HIH-2011-17
Record Dates: First submitted 2013-10-24; First posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Hepatic Injury
Keywords: Acetaminophen; Suicide; Attempts; Early Predictors of Hepatic Injury; Childhood Suicidal Behaviour
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Case-Only
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Biospecimen Retention: Samples Without DNA — The initial and maximum levels of the biochemical parameters will be registered from the electronic biochemistry files of each patient: GLU, basic phosphatase (BP), INR, ALT, and AST.
Oversight: Data Monitoring Committee: No

SUMMARY:
A: Early predictors of hepatic injury after suicide attempt with acetaminophen:

To explore the following in a pediatric population with acetaminophen overdose due to suicide attempt: 1) the prevalence of episodes of pre- and in-hospital vomiting and the relationship between the total number of vomiting episodes and hepatic injury, 2) the relevance of the early initiation of N-acetylcysteine (NAC) treatment to hepatic injury, and 3) the presence/absence of illness prior to the suicide attempt and hepatic injury.

B: Characteristics, social behaviour, trends and risk factors:

1. To explore the relationship between children admitted to a paediatric department as a result of suicide attempts with acetaminophen and their parents and friends. 2. To determine the extent to which the children had attempted to speak to their parents or other adults about their problems before their suicide attempts. 3. To determine the prevalence of self-mutilation among children with suicidal behaviour. 4. To examine the reasons for these suicide attempts.

C: Establishment of the expression of cytochrome P450 in a pediatric including the age-adjusted activities.

Urine samples will be analyzed using an HPLC tandem mass spectrometric method, which we have already established in our lab.

There will be categorized three groups for comparison:

1. An age-appropriate background population (approximately 200 patients)
2. Paediatric patients that have been admitted to Rigshospitalet, due to severe hepatic injury (approximately 50 patients)
3. Other pediatric patients admitted to their local hospital because of acetaminophen poisoning (approximately 200 patients) A control urine sample will be analyzed three months after the suicide attempt.

ELIGIBILITY:
Inclusion Criteria:

* 8-18 years-old, who tried to commit suicide with acetaminophen.
* Children are only included if they have answered all our standard questions.

Exclusion Criteria:

* Children with known liver disease prior to the suicide attempt.
* If a child have several suicide attempts during the inclusion-period, only the 1st will be included.
* Suicide attempts with other agents than acetaminophen.
* Children taking medication that enhance the induction of the cytochrome P450 system, increase the production of toxic metabolites, and aggravate the hepatic injury, such as ethanol, rifampin, isoniazid, barbiturates, and carbamazepine, will be excluded.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric Department, children/adolescents who have tried to commit suicide with acetaminophen (8-18 years-old)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2005-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Early predictors of hepatic injury | 2 years
  1) To identify early clinical and biochemical predictors of hepatoxicity in children and adolescents after the ingestion of a single acetaminophen overdose as a part of a suicide attempt e.g. pre-hospital vomiting, in-hospital vomiting, stomach pains, latency time before NAC treatment, illness prior to the suicide attempt. The initial and maximum levels of the following biochemical parameters are registered from the electronic biochemistry files of each patient: gluthathione (GLU), basic phosphatase (BP), INR, ALT, AST, and s-acetaminophen.

SECONDARY OUTCOMES:
Expression of CYP 1A2 in a pediatric population | 2 years
  The expression of cytochrome P450 in a pediatric population including the age-adjusted activities.
  Urine samples will be analyzed using an HPLC tandem mass spectrometric method, which we have already established in our lab.
  There will be categorized three groups for comparison:
  An age-appropriate background population (approximately 200 patients) Paediatric patients that have been admitted to Rigshospitalet, due to severe hepatic injury (approximately 50 patients) Other pediatric patients admitted to their local hospital because of acetaminophen poisoning (approximately 200 patients) A control urine sample will be analyzed three months after the suicide attempt.
Characteristics, social behaviour, trends and risk factors | 2 years
  1)The relationship children with suicidal behaviour have with their parents and friends. 2)The prevalence of self-mutilation among children with suicidal behaviour. 3)The purposes and main reasons for suicide attempts among children/adolescents. 4) The extent to which these suicide attempts are planned. 5) The extent of acetaminophen intake.

CONTACTS AND LOCATIONS:
Locations (1):
- Nordsjællands Hospital, Hillerød, Denmark